CLINICAL TRIAL: NCT07304791
Title: A Randomized, Single-Blind, Placebo-Controlled, Phase 1 Single Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of BEAM-103 in Healthy Subjects
Brief Title: This is a Phase 1, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of BEAM-103 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: BTX-103-001
Record Dates: First submitted 2025-09-29; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects; Healthy Participant Study
Keywords: ESCAPE; BEAM-103

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BEAM-103 Drug Product (Experimental): BEAM-103 is a monoclonal antibody that will be administered in single dose ascending dose cohorts as an intravenous infusion through the arm.
  Interventions: Drug: BEAM-103
- Placebo (Placebo Comparator): Normal Saline Solution will be administered as a matching place in single dose ascending dose cohorts as an intravenous infusion through the arm.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: BEAM-103 — • BEAM-103 is a monoclonal antibody administered as a single intravenous dose
  Arms: BEAM-103 Drug Product
Drug: Placebo Comparator — • The matching placebo comparator is administered as a single intravenous dose
  Arms: Placebo

SUMMARY:
The purpose of this Phase I single ascending dose study is to evaluate the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of BEAM-103 in healthy subjects between the ages of 18 and 55. The main questions the study aims to answer are:

* Safety and tolerability of BEAM-103
* The pharmacokinetic (PK) profile and pharmacodynamic (PD) characteristics of EAM-103
* The effect of BEAM-103 on hematologic parameters
* To assess the immunogenicity of BEAM-103

Researchers will determine and establish the therapeutic window of the antibody and select optimal doses for future trials in patients.

Subjects will:

* Be asked to participate in the study for a duration of 4-5 months total
* Be asked to sign informed consent
* Be assessed for eligibility
* Provide medical and medication history
* Receive a single intravenous infusion of BEAM-103 or placebo on study Day 1 according to their assigned cohort
* Be followed up to 4 months after infusion

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to ≤55 years
* Body mass index (BMI) of 18.5 to 25 kg/m2
* Morning neutrophil count ≥2.6 × 109 cells/L for Black/African American subjects or ≥3.5 ×109 cells/L for Caucasian/Other subjects
* Baseline hemoglobin value of ≥14 g/dL for males and ≥12 g/dL for females
* Baseline platelet count of >150 × 109/L.
* Subjects must be in general good health without significant medical conditions (based on physical exam, electrocardiogram (ECG), and laboratory test results with no clinically significant deviations), per the investigator's assessment

Exclusion Criteria:

* Known hypersensitivity to any component of the investigational medicinal product (IMP).
* Participation in another clinical trial involving treatment with an investigational agent within 90 days of informed consent is prohibited.
* Positive serum pregnancy test or breastfeeding at screening (female participants).
* Live virus vaccination within 4 weeks prior to signing informed consent.
* Any severe or uncontrolled medical condition (eg. severe asthma or severe peanut allergy) that in the opinion of the investigator would put the subject at undue medical risk or impair the ability to interpret study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-05-29 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of single ascending doses of BEAM-103 | from enrollment to the end of study at 5 months
  Incidence of treatment-emergent AEs, serious AEs, severe AEs, AEs related to BEAM-103

SECONDARY OUTCOMES:
Change in Free Stem Cell Factor (SCF) in Peripheral Blood Over Time | from the start of treatment to the end of study at 5 months
  Concentration of SCF in peripheral blood measured in nanograms per milliliter (mL)
Change in Tryptase Level in Peripheral Blood Over Time | from the start of treatment to the end of study at 5 months
  Serum tryptase concentration measured in nanograms per milliliter (ng/mL)
Change in Reticulocyte Count in Peripheral Blood Over Time | From enrollment to end of study at 5 months
  Absolute reticulocyte count measured in cells per microliter (cells/µL)
Change in Neutrophil Count in Peripheral Blood Over Time | From enrollment to end of study at 5 months
  Absolute neutrophil count measured in cells per microliter (cells/µL)
Maximum Observed Plasma Concentration (Cmax) | From enrollment to end of study at 5 months
  Cmax will be calculated as the highest observed plasma/blood/serum concentration following drug administration
Area Under the Plasma Concentration-Time Curve to Last Quantifiable Concentration (AUClast) | From enrollment to end of study at 5 months
  AUClast will be calculated from time zero to the time of the last quantifiable concentration
Area Under the Plasma Concentration-Time Curve to Infinity (AUC∞) | From enrollment to end of study at 5 months
  AUC∞ will be calculated as AUClast plus Clast divided by λz
Terminal Elimination Half-Life (t½) | From enrollment to end of study at 5 months
  t½ will be estimated from the terminal elimination phase of the plasma concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Study Site, London, United Kingdom